CLINICAL TRIAL: NCT06123221
Title: COMPARISON OF IMPLANT INSTALLATION USING THE TRANSCRESTAL APPROACH WITH OSSEODENSIFICATION OR THE LATERAL WINDOW TECHNIQUE WITH SINUS LIFT: A RANDOMIZED CONTROLLED TRIAL.
Brief Title: SINUS FLOOR WITH OSSEODENSIFICATION OR LATERAL WINDOW
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Alex Nogueira Haas, Professor, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UFRGS-Cuiaba
Record Dates: First submitted 2022-11-23; First posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2022-11

CONDITIONS: Sinus Tract; Dental Implant Failed

STUDY DESIGN:
Intervention Model Description: Parallel randomized controlled trial
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Osseodensification (Experimental): Sinus floor elevation with osseodensification and concomitant implant installation
  Interventions: Procedure: Osseodensification with Versah system
- Lateral window (Active Comparator): Sinus floor elevation with lateral window and concomitant implant installation
  Interventions: Procedure: Lateral window

INTERVENTIONS:
Procedure: Osseodensification with Versah system — Access to the bone crest will be performed through a slightly palatinized crestal incision, and a full-thickness mucoperiosteal flap will be elevated. Implant site preparation will be performed according to the bone densification drilling sequence established by the Densah® technique protocol
  Arms: Osseodensification
Procedure: Lateral window — A full-thickness mucoperiosteal flap will be elevated. The lateral window will be made with a spherical diamond drill (number 8) at 20,000 rpm. The mesiodistal and apicocoronal dimensions of the lateral access window to the sinus will be measured in all the participants using a caliper. Sinus membrane elevation will be performed with manual instruments.
  Arms: Lateral window

SUMMARY:
This study will compare patient-reported outcomes, as well as the type and incidence of complications, and bone marginal loss after 12 months in implants installed using the transcrestal approach (tSFE) with an osseodensification system (performed according to the protocol by Huwais et al. 2018), or installed simultaneously using the lateral window technique (lSFE) with sinus lift. A blind, randomized, controlled clinical trial will be carried out with individuals over 18 years old, and with single tooth loss in the posterior maxilla, where the residual bone height (RBH) is 3 to 5 mm. The tSFE will be performed with osseodensification burs (Densa Bur, Versah, USA) using a counterclockwise motion, associated to synthetic biomaterial (hydroxyapatite and beta-tricalcium phosphate). The lSFE technique will require the sinus to be filled with the same biomaterial as the group using the other technique, and the antrostomy to be covered with a polydioxanone-based membrane. The patient's post-operatory perceptions will be evaluated by self-administered questionnaires quantifying social and professional isolation, physical appearance, duration and changes in quality of life, eating and speech, diet variations, and sleep deficiency for 2 weeks after the procedure. Pain will be assessed with the visual analogue scale (VAS). Immediately after prosthetic rehabilitation, cone beam tomography will be performed. Controls at 6 and 12 months will be performed. In these images, the marginal bone level in relation to a fixed reference point on the implants (upper part of the platform) will be measured mesially and distally in each implant, using a specific program (ImageJ - version 1.49v / NIH software - Bethesda, MD, USA). Generalized estimating equations will be used to compare the two treatments overtime. The significance level used will be 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Maxillary sinuses that have residual bone height between at least 3 mm and 5 mm;
* Width of the residual bone ridge that allows the insertion of an implant with a diameter of 4 mm;
* Tomographic thickness of Schneider's membrane with a maximum of 5 mm in the region to be operated;
* Residual ridge with ≥2 mm of medullary bone in the bucco-palatal direction, with a 1/1 ratio of medullary and cortical bone to achieve predictable plastic expansion;
* Patients with adequate interarch space for placement of the prosthetic crown;
* Good physical health status (ASA1 and ASA2, according to the Physical Status Classification System - American Society of Anesthesiologists);
* At least 6 months since the last tooth loss in the region to be operated;

Exclusion Criteria:

* - Those with sinus pathology;
* Heavy smokers (more than 10 cigarettes a day);
* Those with a history of head and neck radiotherapy;
* Those who have already undergone bone augmentation in any of the targeted surgical areas;
* Immunodeficiency of any nature;
* Emotional instability and psychiatric problems;
* Pregnancy;
* Current use of oral bisphosphonates or history of using injectable bisphosphonate;
* Patients with active periodontitis defined by the presence of subgingival bleeding greater than 10%;
* Documented allergy to drugs or dental materials involved in the experimental protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Pain level | baseline
  visual analogue scale (VAS), ranging from "0 - no pain" to "100 - worst imaginable pain"
Pain level | day 1
  visual analogue scale (VAS), ranging from "0 - no pain" to "100 - worst
Pain level | day 2
  visual analogue scale (VAS), ranging from "0 - no pain" to "100 - worst
Pain level | day 3
  visual analogue scale (VAS), ranging from "0 - no pain" to "100 - worst
Pain level | day 4
  visual analogue scale (VAS), ranging from "0 - no pain" to "100 - worst
Pain level | day 7
  visual analogue scale (VAS), ranging from "0 - no pain" to "100 - worst
Pain level | day 14
  visual analogue scale (VAS), ranging from "0 - no pain" to "100 - worst

SECONDARY OUTCOMES:
Medication Diary (number of doses of Ibuprofen 600mg) | baseline
  Rescue anti-inflammatory drug dosage (i.e. number of ibuprofen 600 mg tablets), and name of other types of drugs taken as of the day of surgery up to the 14th postoperative day, recorded daily in a medication diary
Medication Diary (number of doses of Ibuprofen 600mg) | day 1
  Rescue anti-inflammatory drug dosage (i.e. number of ibuprofen 600 mg tablets), and name of other types of drugs taken as of the day of surgery up to the 14th postoperative day, recorded daily in a medication diary
Medication Diary (number of doses of Ibuprofen 600mg) | day 2
  Rescue anti-inflammatory drug dosage (i.e. number of ibuprofen 600 mg tablets), and name of other types of drugs taken as of the day of surgery up to the 14th postoperative day, recorded daily in a medication diary
Medication Diary (number of doses of Ibuprofen 600mg) | day 3
  Rescue anti-inflammatory drug dosage (i.e. number of ibuprofen 600 mg tablets), and name of other types of drugs taken as of the day of surgery up to the 14th postoperative day, recorded daily in a medication diary
Medication Diary (number of doses of Ibuprofen 600mg) | day 4
  Rescue anti-inflammatory drug dosage (i.e. number of ibuprofen 600 mg tablets), and name of other types of drugs taken as of the day of surgery up to the 14th postoperative day, recorded daily in a medication diary
Medication Diary (number of doses of Ibuprofen 600mg) | day 5
  Rescue anti-inflammatory drug dosage (i.e. number of ibuprofen 600 mg tablets), and name of other types of drugs taken as of the day of surgery up to the 14th postoperative day, recorded daily in a medication diary
Medication Diary (number of doses of Ibuprofen 600mg) | day 6
  Rescue anti-inflammatory drug dosage (i.e. number of ibuprofen 600 mg tablets), and name of other types of drugs taken as of the day of surgery up to the 14th postoperative day, recorded daily in a medication diary
Medication Diary (number of doses of Ibuprofen 600mg) | day 7
  Rescue anti-inflammatory drug dosage (i.e. number of ibuprofen 600 mg tablets), and name of other types of drugs taken as of the day of surgery up to the 14th postoperative day, recorded daily in a medication diary
Medication Diary (number of doses of Ibuprofen 600mg) | day 8
  Rescue anti-inflammatory drug dosage (i.e. number of ibuprofen 600 mg tablets), and name of other types of drugs taken as of the day of surgery up to the 14th postoperative day, recorded daily in a medication diary
Medication Diary (number of doses of Ibuprofen 600mg) | day 9
  Rescue anti-inflammatory drug dosage (i.e. number of ibuprofen 600 mg tablets), and name of other types of drugs taken as of the day of surgery up to the 14th postoperative day, recorded daily in a medication diary
Medication Diary (number of doses of Ibuprofen 600mg) | day 10
  Rescue anti-inflammatory drug dosage (i.e. number of ibuprofen 600 mg tablets), and name of other types of drugs taken as of the day of surgery up to the 14th postoperative day, recorded daily in a medication diary
Medication Diary (number of doses of Ibuprofen 600mg) | day 11
  Rescue anti-inflammatory drug dosage (i.e. number of ibuprofen 600 mg tablets), and name of other types of drugs taken as of the day of surgery up to the 14th postoperative day, recorded daily in a medication diary
Medication Diary (number of doses of Ibuprofen 600mg) | day 12
  Rescue anti-inflammatory drug dosage (i.e. number of ibuprofen 600 mg tablets), and name of other types of drugs taken as of the day of surgery up to the 14th postoperative day, recorded daily in a medication diary
Medication Diary (number of doses of Ibuprofen 600mg) | day 13
  Rescue anti-inflammatory drug dosage (i.e. number of ibuprofen 600 mg tablets), and name of other types of drugs taken as of the day of surgery up to the 14th postoperative day, recorded daily in a medication diary
Medication Diary (number of doses of Ibuprofen 600mg) | day 14
  Rescue anti-inflammatory drug dosage (i.e. number of ibuprofen 600 mg tablets), and name of other types of drugs taken as of the day of surgery up to the 14th postoperative day, recorded daily in a medication diary

OTHER OUTCOMES:
Level of discomfort | as recorded on day 0 (night), +1, +2, +3, +4, +7, and +14,
  Level of discomfort as recorded on a 5-point rating scale ranging from "no discomfort"; "little discomfort"; "discomfort"; "a lot of discomfort" and "very high discomfort"
Limitations in daily functions | as recorded on day 0 (night), +1, +2, +3, +4, +7 and + 14
  Limitations in daily functions (i.e. swallowing, breathing, continuing daily activities, eating, speaking, opening the mouth), on a 5-point rating scale ranging from "no limitations" to "unable to eat all kinds of food" (for the item "eat"), and from "no difficulty" to "extreme difficulty" (for the other items );
Incidence of postoperative signs and symptoms | day 0 (night), +1, +2, +3, +4, +7 and +14;
  Incidence of swelling, nausea, bruising, nasal discharge/bleeding, nasal stuffiness, bad taste/smell
Willingness to undergo the same type of surgery | recorded on day +14
  a 4-point rating scale ranging from "no problem to repeat surgery if needed" to "I will never have this type of surgery again."
Clinical Outcomes | 7 and 14 days after surgery
  Membrane perforation (yes or no) will be evaluated during the transoperative period. In addition, the following clinical outcomes will be evaluated: Face edema (yes or no);
  * Facial hematoma (yes or no);
  * Presence of suppuration;
  * Suture dehiscence.
Cinical evaluation of Implant failure | through study completion, an average of 18 months
  Implant loss may occur during the phase of osseointegration (early) or at a later time when the previously achieved osseointegration is lost (late). Implant loss defined by lack of osseointegration represented by mobility, and will be assessed at throughout the entire search
Peri-implant clinical examinations | 1 and 12 months after the installation of the prosthesis
  probing depth in millimeters will be evaluated at six sites per implant (mesiobuccal, buccal, distobuccal, and mesiolingual/palatal, lingual/palatal, distolingual/palatal).
Peri-implant clinical examinations | 1 and 12 months after the installation of the prosthesis
  submucosal bleeding points after probing will be evaluated at six sites per implant (mesiobuccal, buccal, distobuccal, and mesiolingual/palatal, lingual/palatal, distolingual/palatal).
Tomographic outcomes | 1 and 12 months after the installation of the prosthesis
  The images will be used to measure the marginal bone level mesially and distally in each implant, in relation to a fixed reference point on the implants (upper part of the platform), using a specific program (ImageJ)

CONTACTS AND LOCATIONS:
Locations (1):
- Alex Haas, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Background] Farina R, Franceschetti G, Travaglini D, Consolo U, Minenna L, Schincaglia GP, Riccardi O, Bandieri A, Maietti E, Trombelli L. Morbidity following transcrestal and lateral sinus floor elevation: A randomized trial. J Clin Periodontol. 2018 Sep;45(9):1128-1139. doi: 10.1111/jcpe.12985. Epub 2018 Aug 3. PMID 29992594
- [Result] Huwais S, Mazor Z, Ioannou AL, Gluckman H, Neiva R. A Multicenter Retrospective Clinical Study with Up-to-5-Year Follow-up Utilizing a Method that Enhances Bone Density and Allows for Transcrestal Sinus Augmentation Through Compaction Grafting. Int J Oral Maxillofac Implants. 2018 Nov/Dec;33(6):1305-1311. doi: 10.11607/jomi.6770. PMID 30427961
- [Result] Starch-Jensen T, Jensen JD. Maxillary Sinus Floor Augmentation: a Review of Selected Treatment Modalities. J Oral Maxillofac Res. 2017 Sep 30;8(3):e3. doi: 10.5037/jomr.2017.8303. eCollection 2017 Jul-Sep. PMID 29142655
- [Result] Franceschetti G, Rizzi A, Minenna L, Pramstraller M, Trombelli L, Farina R. Patient-reported outcomes of implant placement performed concomitantly with transcrestal sinus floor elevation or entirely in native bone. Clin Oral Implants Res. 2017 Feb;28(2):156-162. doi: 10.1111/clr.12774. Epub 2016 Jan 8. PMID 26749535
- [Result] Bacevic M, Compeyron Y, Lecloux G, Rompen E, Lambert F. Intraoperative and postoperative outcomes of sinus floor elevation using the lateral window technique versus the hydrodynamic transalveolar approach: a preliminary randomized controlled trial. Clin Oral Investig. 2021 Sep;25(9):5391-5401. doi: 10.1007/s00784-021-03847-2. Epub 2021 Mar 10. PMID 33694027
- [Result] Starch-Jensen T, Bruun NH. Patient's perception of recovery after osteotome-mediated sinus floor elevation with Bio-Oss collagen compared with no grafting material: a randomized single-blinded controlled trial. Int J Implant Dent. 2021 Mar 22;7(1):20. doi: 10.1186/s40729-021-00302-5. PMID 33748923
- [Result] Pikos MA, Miron RJ. To Drill or to Densify? Clinical Indications for the Use of Osseodensification. Compend Contin Educ Dent. 2019 May;40(5):276-281; quiz 282. PMID 31067068
- [Result] Huwais S, Meyer EG. A Novel Osseous Densification Approach in Implant Osteotomy Preparation to Increase Biomechanical Primary Stability, Bone Mineral Density, and Bone-to-Implant Contact. Int J Oral Maxillofac Implants. 2017 Jan/Feb;32(1):27-36. doi: 10.11607/jomi.4817. Epub 2016 Oct 14. PMID 27741329